CLINICAL TRIAL: NCT03064373
Title: Mother to Newborn Transmission of Staphylococcus Aureus and the Dynamics of S. Aureus Carriage During the First Years of Life
Brief Title: Mother to Newborn Transmission of Staphylococcus Aureus and Dynamics of S.Aureus Carriage During the First Years Life
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: The Israel Science Foundation (Unknown)
Responsible Party: Principal Investigator, Gili Regev-Yochay MD, Director, Infection Control Unit, Sheba Medical Center
Other Study IDs: 5534-08
Record Dates: First submitted 2017-02-22; First posted 2017-02-27 (Actual); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Staphylococcus Aureus
Keywords: S. aureus; carriage; mother-neonatal transmission; microbiome
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — S. aureus and S. pneumoniae
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Staphylococcus aureus (SA) is a significant cause of community and hospital acquired infections. SA is carried by approximately 30% of healthy adults. Similar carriage rates have been reported in very young infants and newborns. Previous studies have suggested that the source of SA carriage in young children is SA carried by their mothers. Possible modes of transmission from mother to child are transmission during passage through a colonized birth canal, through lactation and/or close contact.

We aim to 1) Define the route of transmission between mother and newborn. 2) Assess the dynamics of S. aureus carriage during the first years of life and specifically determine risk factors for becoming a persistent carrier of S. aureus

DETAILED DESCRIPTION:
Design:

prospective cohort study which will examine the risk of exposure to S. aureus carrier mother on the outcome: S. aureus carriage by newborns following delivery and at discharge.

1. Risk of vertical transmission during delivery will be assessed by comparing a cohort of newborns to vaginal S. aureus carrier mothers to a cohort of newborns of mothers not carrying S. aureus vaginally.
2. Risk of horizontal transmission during the first days of life will be assessed by following a cohort of newborns not colonized on delivery day. The main exposure of interest is maternal nasal SA carriage.Target populations: 300 mother - newborn pairs.

Setting:

Sheba Medical Center obstetrical unit and nursery Gravid women will be recruited during antenatal visit at the Sheba medical Center, 1-4 weeks prior to labor. Women who will agree to participate and sign an informed consent will be screened for nasal and vaginal carriage of S. aureus. Newborns will be screened on delivery day and on discharge day.

Inclusion criteria:

1. Gravid women expected to deliver within 4 weeks.
2. Women who agree to participate and sign an informed consent
3. Women who are S. aureus carriers at the time of recruit.

Exclusion criteria:

1. Prolonged (>6 days) newborn hospitalization.
2. Women who did not give birth eventually at the Sheba Medical Center.
3. Women who's newborns were not screened at least once during delivery hospitalization.

Enrollment:

300 consecutive women who are defined as S. aureus carriers (see definitions below).

Screening will include:

Stage I before discharge:

1. Women - nasal screenings:

   A) On recruitment day (~1-4 weeks before labor), B) During hospitalization for delivery. Vaginal screening will be performed during the routine gynecologic examination on delivery day.
2. Newborns - will be screened A) On birth day, at entrance to the nursery. B) On discharge day. Screening will include nasal nares, umbilical, ear and rectal swabbing on each screening while hospitalized.
3. Data collection by questionnaires filled by recruited women.
4. Data collection from medical files of the maternity ward.

Stage II after discharge until age 5 years:

1. Mothers - monthly nasal swab for 12 months.
2. Children - monthly nasal, nasopharyngeal and rectal swabs for 12 months.
3. Same screen annually until the child is 5years old.
4. Data collection by questionnaires filled by the mothers.

ELIGIBILITY:
Inclusion Criteria:

1. Gravid women expected to deliver within 4 weeks.
2. Women who agree to participate and sign an informed consent
3. Women who are S. aureus carriers at the time of recruit.

Exclusion Criteria:

1. Prolonged (>6 days) newborn hospitalization.
2. Women who did not give birth eventually at the Sheba Medical Center.
3. Women who's newborns were not screened at least once during delivery hospitalization.

Enrollment:

300 consecutive women who are defined as S. aureus carriers (see definitions below).

Ages: 24 Hours to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 300 mother - newborn pairs.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2008-12-17 (Actual); Primary Completion 2022-12-17 (Estimated); Study Completion 2023-06-17 (Estimated)

PRIMARY OUTCOMES:
S. aureus carriage | 5 years
  Carriage of S. aurues in any of the sites

CONTACTS AND LOCATIONS:
Overall Officials: Dror Charats, Prof., Study Chair — IRB Committee.Sheba Medical Center Israel
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leshem E, Maayan-Metzger A, Rahav G, Dolitzki M, Kuint J, Roytman Y, Goral A, Novikov I, Fluss R, Keller N, Regev-Yochay G. Transmission of Staphylococcus aureus from mothers to newborns. Pediatr Infect Dis J. 2012 Apr;31(4):360-3. doi: 10.1097/INF.0b013e318244020e. PMID 22189535